CLINICAL TRIAL: NCT01736085
Title: Distribution of Voucher vs. Direct Mailing of Nicotine Patches to Quitline Smokers
Brief Title: Providing Free Nicotine Patches to Quitline Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P121218
Record Dates: First submitted 2012-11-15; First posted 2012-11-29 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: tobacco cessation; smoking cessation; nicotine; telephone counseling; self-help; smoking abstinence; tobacco use disorder; nicotine replacement therapy; voucher
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Material Group (No Intervention): Subjects will receive self-help materials
- Materials plus Voucher (Active Comparator): Subjects will receive self-help materials and a voucher for 2 week's worth of nicotine patches
  Interventions: Behavioral: Voucher
- Materials plus Patches (Active Comparator): Subjects will receive self-help materials and a 2 week's worth of nicotine patches
  Interventions: Drug: Nicotine patches
- Counseling (Active Comparator): Subjects will receive up to 5 sessions of telephone counseling
  Interventions: Behavioral: Telephone counseling
- Counseling plus Voucher (Active Comparator): Subjects will receive up to 5 sessions of telephone counseling plus a voucher for 2 week's worth of nicotine patches.
  Interventions: Behavioral: Telephone counseling; Behavioral: Voucher
- Counseling plus Patches (Active Comparator): Subjects will receive up to 5 sessions of telephone counseling plus 2 week's worth of nicotine patches.
  Interventions: Behavioral: Telephone counseling; Drug: Nicotine patches

INTERVENTIONS:
Behavioral: Telephone counseling — Telephone counseling is conducted in the appropriate language (English and Spanish) by veteran counselors at the California Smokers' Helpline. Subjects will receive free proactive telephone counseling to help them set up quit smoking plans. The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. It includes a 30-minute comprehensive pre-quit session (motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four 10-minute proactive follow-up calls. The counseling protocol has several distinguishing features: proactive follow-up counseling calls, a manualized (i.e., semi-structured) protocol and relapse-sensitive scheduling
  Arms: Counseling; Counseling plus Patches; Counseling plus Voucher
Behavioral: Voucher — Subjects will receive a voucher for nicotine patches.
  Subjects randomized into the voucher condition will receive a voucher that can be exchanged for two weeks' worth of free starter kit nicotine patches by calling a dedicated phone number (Quit Boost). The voucher will be mailed the day after the screening intake. Subjects who smoke 11 or more cigarettes per day will receive 21 mg patches; smoke 10 or less per day will receive 14 mg patches. Subjects will be encouraged to start using these patches on their quit date.
  Other Names: Voucher for nicotine patch
  Arms: Counseling plus Voucher; Materials plus Voucher
Drug: Nicotine patches — Subjects will receive nicotine patches directly sent to their home. Subjects randomized into the patch condition will receive two weeks' worth of free starter kit nicotine patches directly. The patches will be mailed directly to their home the day after screening intake. Subjects who smoke 11 or more cigarettes per day will receive 21 mg patches; smoke 10 or less per day will receive 14 mg patches. Subjects will be encouraged to start using these patches on their quit date.
  Other Names: Nicotine patches sent directly
  Arms: Counseling plus Patches; Materials plus Patches

SUMMARY:
The California Smokers' Helpline will conduct a 3 X 2 (nicotine patch by counseling condition) randomized trial to test the provision of nicotine patches to help smokers calling a telephone quitline. The study assesses one factor related to nicotine patches with 3 levels: sending patches directly from the Helpline, providing vouchers that can be redeemed for patches, and usual care. A second factor is counseling plus materials versus materials only. This proposed study has the following specific aims:

1. To demonstrate that a voucher for free nicotine patches will increase the quit rate for smokers who do not have access to free nicotine replacement therapy (NRT)
2. To demonstrate that sending patches directly from a quitline would outperform sending vouchers for free NRT, since the vouchers impose an additional barrier to those who want to quit
3. To determine the effect of telephone counseling in the context of nicotine patch distribution and if any interaction effects exist between counseling and patch conditions

DETAILED DESCRIPTION:
Tobacco smoking leads to nicotine dependence and serious health consequences. Telephone counseling has been shown to improve smokers' chances of quitting and is the most accessible of the three evidence-based forms of counseling (individual face-to-face, group, and telephone). It is well established that offering free NRT can attract many more smokers to call a quitline. However, how much the offer of free NRT helps quitline callers quit successfully is less well documented. There is currently no consistent guideline for quitline practice. We want to determine whether two weeks' worth of starter kit nicotine patches is efficacious for smokers who don't have access to free nicotine patches or quitting aids. The study also will provide data regarding the impact of a barrier to obtaining quitting aids by contrasting a direct mailing condition with a voucher condition. Further, the study will help us determine the effect of telephone counseling in the context of nicotine patch distribution and if any interaction effects exist between counseling and patch conditions

The study uses a randomized controlled design. Smokers who call the Helpline during the recruitment phase, who meet eligibility requirements for the trial and give consent will be randomly assigned to one of six groups along two factors (nicotine patch and telephone counseling), as described below.

The 6 randomized groups are as follows: Group 1: Materials, Group 2: Voucher + Materials, Group 3: Patches + Materials, Group 4: Counseling, Group 5: Voucher + Counseling, Group 6: Patches + Counseling

Two months and seven months after their initial contact with the Helpline, all participants will receive two Assessment Interviews by phone. The interview will cover, as appropriate, smoking status, use of nicotine patches and other quitting aids, history of quitting, and satisfaction with services provided. The Assessment Interview lasts from 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Current smoker
* First time quitline caller
* Not eligible for nicotine patches through other programs such as MediCal or Los Angeles County which provides free nicotine patches
* English and/or Spanish speaking
* Valid phone number
* Valid address
* CA resident
* Gave consent to participate in study and evaluation

Exclusion Criteria:

* Contraindication(s) to nicotine patches
* Uses a form of tobacco other than cigarettes
* Plans to use Chantix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3706 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego; California Smokers' Helpline, San Diego, California, United States

REFERENCES:
- [Background] Zhu SH, Anderson CM, Tedeschi GJ, Rosbrook B, Johnson CE, Byrd M, Gutierrez-Terrell E. Evidence of real-world effectiveness of a telephone quitline for smokers. N Engl J Med. 2002 Oct 3;347(14):1087-93. doi: 10.1056/NEJMsa020660. PMID 12362011
- [Background] Anderson CM, Zhu SH. Tobacco quitlines: looking back and looking ahead. Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i81-6. doi: 10.1136/tc.2007.020701. PMID 18048638
- [Background] Cummings KM, Fix BV, Celestino P, Hyland A, Mahoney M, Ossip DJ, Bauer U. Does the number of free nicotine patches given to smokers calling a quitline influence quit rates: results from a quasi-experimental study. BMC Public Health. 2010 Apr 7;10:181. doi: 10.1186/1471-2458-10-181. PMID 20374628
- See also: California Smokers' Helpline, University of California, San Diego — http://www.californiasmokershelpline.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Materials Plus Voucher: Subjects will receive self-help materials and a voucher for 2 week's worth of nicotine patches
  Voucher: Subjects will receive a voucher for nicotine patches.
  Subjects randomized into the voucher condition will receive a voucher that can be exchanged for two weeks' worth of free starter kit nicotine patches by calling a dedicated phone number (Quit Boost). The voucher will be mailed the day after the screening intake. Subjects who smoke 11 or more cigarettes per day will receive 21 mg patches; smoke 10 or less per day will receive 14 mg patches. Subjects will be encouraged to start using these patches on their quit date.
- Materials Plus Patches: Subjects will receive self-help materials and a 2 week's worth of nicotine patches
  Nicotine patches: Subjects will receive nicotine patches directly sent to their home.
  Subjects randomized into the patch condition will receive two weeks' worth of free starter kit nicotine patches directly. The patches will be mailed directly to their home the day after screening intake. Subjects who smoke 11 or more cigarettes per day will receive 21 mg patches; smoke 10 or less per day will receive 14 mg patches. Subjects will be encouraged to start using these patches on their quit date.
- Counseling: Subjects will receive up to 5 sessions of telephone counseling
  Telephone counseling: Telephone counseling is conducted in the appropriate language (English and Spanish) by counselors at the California Smokers' Helpline. Subjects will receive free proactive telephone counseling to help them set up quit smoking plans. The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. It includes a 30-minute comprehensive pre-quit session (motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four 10-minute proactive follow-up calls. The counseling protocol has several distinguishing features: proactive follow-up counseling calls, a manualized (i.e., semi-structured) protocol and relapse-sensitive scheduling
- Counseling Plus Voucher: Subjects will receive up to 5 sessions of telephone counseling plus a voucher for 2 week's worth of nicotine patches.
  Telephone counseling: Telephone counseling is conducted in the appropriate language (English and Spanish) by counselors at the California Smokers' Helpline. Subjects will receive free proactive telephone counseling to help them set up quit smoking plans. The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. It includes a 30-minute comprehensive pre-quit session (motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four 10-minute proactive follow-up calls. The counseling protocol has several distinguishing features: proactive follow-up counseling calls, a manualized (i.e., semi-structured) protocol and relapse-sensitive scheduling
  Voucher: Subjects will receive a voucher for nicotine patches.
  Subjects ra
- Counseling Plus Patches: Subjects will receive up to 5 sessions of telephone counseling plus 2 week's worth of nicotine patches.
  Telephone counseling: Telephone counseling is conducted in the appropriate language (English and Spanish) by counselors at the California Smokers' Helpline. Subjects will receive free proactive telephone counseling to help them set up quit smoking plans. The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. It includes a 30-minute comprehensive pre-quit session (motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four 10-minute proactive follow-up calls. The counseling protocol has several distinguishing features: proactive follow-up counseling calls, a manualized (i.e., semi-structured) protocol and relapse-sensitive scheduling
  Nicotine patches: Subjects will receive nicotine patches directly sent to their home.
  Subj
Period: Overall Study
Arm/Group | Material Group | Materials Plus Voucher | Materials Plus Patches | Counseling | Counseling Plus Voucher | Counseling Plus Patches
Started | 529 | 530 | 793 | 530 | 530 | 794
Completed | 529 | 530 | 793 | 530 | 530 | 794
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Material Group | Materials Plus Voucher | Materials Plus Patches | Counseling | Counseling Plus Voucher | Counseling Plus Patches | Total
Number analyzed (Participants) | 529 | 530 | 793 | 530 | 530 | 794 | 3706
Age, Customized [Count of Participants; unit: Participants] — Population: 2 people dropped per subjects' request (materials only and patches + materials)
  Participants
    18-24 years | 55 | 70 | 77 | 62 | 52 | 76 | 392
    25-44 years | 203 | 207 | 304 | 211 | 200 | 297 | 1422
    45-64 years | 236 | 217 | 354 | 231 | 245 | 368 | 1651
    65+ years | 35 | 36 | 58 | 26 | 33 | 53 | 241
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 people dropped per subjects' request (materials only and patches + materials)
  Participants
    Female | 279 | 283 | 377 | 244 | 265 | 419 | 1867
    Male | 250 | 247 | 416 | 286 | 265 | 375 | 1839
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 288 | 263 | 438 | 301 | 300 | 465 | 2055
  Black | 70 | 80 | 117 | 59 | 57 | 110 | 493
  Hispanic | 109 | 94 | 140 | 94 | 122 | 139 | 698
  Asian | 15 | 22 | 30 | 21 | 9 | 16 | 113
  American Indian and Alaska Native | 6 | 11 | 12 | 8 | 9 | 10 | 56
  Multi-Race | 39 | 55 | 52 | 41 | 31 | 51 | 269
  Other | 2 | 5 | 4 | 6 | 2 | 3 | 22
Education [Count of Participants; unit: Participants]
  <=12 | 111 | 99 | 132 | 96 | 99 | 123 | 660
  GED/HSD | 150 | 148 | 259 | 159 | 152 | 232 | 1100
  Some College | 218 | 242 | 323 | 222 | 227 | 339 | 1571
  BS/BA + | 50 | 41 | 79 | 53 | 52 | 100 | 375
Cigs per day [Count of Participants; unit: Participants]
  <15 | 223 | 261 | 348 | 201 | 215 | 330 | 1578
  <=15 | 306 | 269 | 445 | 329 | 315 | 464 | 2128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Six Months Prolonged Abstinence
Description: At seven months post enrollment we will conduct a brief telephone survey to assess smoking status. The information obtained will allow us to determine six month prolonged abstinence rates.
Time Frame: Seven months post enrollment
Population: intent-to-treat; we are looking at the marginal means
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: no provision of free nicotine replacement therapy (NRT)
- Voucher: Free nicotine replacement through a voucher system
- Patches: nicotine replacement sent directly
Arm/Group | Usual Care | Voucher | Patches
Number analyzed (Participants) | 1059 | 1060 | 1587
Participants | 61 | 76 | 151

2. Secondary Outcome: Percentage of Smokers Making a 24-hour Quit Attempt
Description: At the follow up evaluation, subjects will be asked if they have made a quit attempt that lasted at least 24 hours.
Time Frame: Two months post enrollment
Population: those evaluated at 2-months; we are looking at the marginal means
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Voucher | Patches
Number analyzed (Participants) | 766 | 802 | 1212
Participants | 455 | 533 | 879

ADVERSE EVENTS:
Arm/Group | Material Group | Materials Plus Voucher | Materials Plus Patches | Counseling | Counseling Plus Voucher | Counseling Plus Patches
Serious Adverse Events (participants affected / at risk) | 0/529 | 0/530 | 0/793 | 0/530 | 0/530 | 0/794
Other Adverse Events (participants affected / at risk) | 0/529 | 0/530 | 0/793 | 0/530 | 0/530 | 0/794

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No